CLINICAL TRIAL: NCT01456052
Title: Phase 2 Assessment of the Relationship Between Serotonin and Efficacy in Ulcerative Colitis: A Multi-Center Randomized, Double Blind, Placebo-Controlled, Pilot Study to Evaluate Safety and Preliminary Efficacy of Orally Administered LX1606 in Subjects With Acute, Mild to Moderate Ulcerative Colitis
Brief Title: A Study to Evaluate Safety and Efficacy of Telotristat Etiprate (LX1606) in Participants With Acute, Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX1606.1-204-UC; LX1606.204 (Other: Lexicon Pharmaceuticals, Inc.); LX1032 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — telotristat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose Telotristat Etiprate (Experimental): 500 mg telotristat etiprate (LX1606) administered orally once daily (QD).
  Interventions: Drug: Telotristat Etiprate
- High Dose Telotristat Etiprate (Experimental): 500 mg telotristat etiprate (LX1606) administered orally three times daily (TID).
  Interventions: Drug: Telotristat Etiprate
- Placebo (Placebo Comparator): Matching placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telotristat Etiprate — 500 mg telotristat etiprate (LX1606) administered orally.
  Arms: High Dose Telotristat Etiprate; Low Dose Telotristat Etiprate
Drug: Placebo — Matching placebo administered orally.
  Arms: Placebo

SUMMARY:
This is a multicenter, placebo-controlled, parallel-group, pilot study to evaluate safety and preliminary effectiveness of two blinded dose levels of telotristat etiprate (LX1606) in participants with acute, mild to moderate ulcerative colitis on 5-aminosalicylic acid/mesalamine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis of at least 6 months duration
* Disease extends at least 15 cm proximally from the anal verge, documented within the past 3 years
* Flare occurs on 5-aminosalicylic acid (5-ASA)/mesalamine therapy and subject is willing to remain on a stable dose for the duration of the study
* Age ≥18 and <70 years of age
* Able and willing to provide written informed consent

Exclusion Criteria:

* Prior terminal ileum or colonic surgery, except appendectomy or hemorrhoid surgery
* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's disease
* Clinical signs of fulminant colitis or toxic megacolon
* History of dysplasia associated lesion or mass (DALM)
* Subjects who have had surgery for ulcerative colitis, or in the opinion of the investigator, are likely to require surgery for ulcerative colitis during the study
* History of primary sclerosing cholangitis
* Any physical or laboratory abnormality deemed by the investigator as clinically significant
* Major surgery within 60 days of Screening
* Use of any investigational agent within 30 days of Screening or any therapeutic protein or antibody within 90 days of Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2013-09-03 (Actual); Study Completion 2013-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Fleming, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (22):
- United States (11):
  - Lexicon Investigational Site, Little Rock, Arkansas
  - Lexicon Investigational Site, Anaheim, California
  - Lexicon Investigational Site, Santa Monica, California
  - Lexicon Investigational Site, Great Neck, New York
  - Lexicon Investigational Site, New York, New York
  - Lexicon Investigational Site, Tulsa, Oklahoma
  - Lexicon Investigational Site, Houston, Texas
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Ogden, Utah
  - Lexicon Investigational Site, Sandy City, Utah
  - Lexicon Investigational Site, Seattle, Washington
- Lithuania (4):
  - Lexicon Investigational Site, Kaunas
  - Lexicon Investigational Site, Klaipėda
  - Lexicon Investigational Site, Šiauliai
  - Lexicon Investigational Site, Vilnius
- Poland (5):
  - Lexicon Investigational Site, Krakow
  - Lexicon Investigational Site, Lodz
  - Lexicon Investigational Site, Sopot
  - Lexicon Investigational Site, Warsaw
  - Lexicon Investigational Site, Wroclaw
- Slovakia (2):
  - Lexicon Investigational Site, Nitra
  - Lexicon Investigational Site, Nové Mesto nad Váhom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 60 participants were to be enrolled and treated in the blinded Treatment period across 24 US and international sites. The recruitment period lasted approximately 10 months.
Pre-assignment Details: The study consisted of an approximately 15 days Screening period prior to the blinded Treatment period.
Period: Overall Study
Arm/Group | Placebo | Low Dose Telotristat Etiprate | High Dose Telotristat Etiprate
Started | 10 | 25 (One subject did not receive any study drug. That subject is not included in the safety population.) | 24
Completed | 8 | 20 | 19
Not Completed | 2 | 5 | 5
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Consent withdrawn | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Treatment Failure | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the safety population. One subject was excluded from the safety population as they did not receive any doses of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Telotristat Etiprate | High Dose Telotristat Etiprate | Total
Number analyzed (Participants) | 10 | 24 | 24 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (16.16) | 45.5 (12.49) | 41.7 (12.69) | 42.8 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 7 | 23
  Male | 6 | 12 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 24 | 22 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Treatment Emergent Adverse Event
Time Frame: 8 weeks
Population: Safety population included all treated participants who had taken any fraction of a study drug dose.
Measure: Number; unit: participants
Groups:
- Low Dose LX1606: 500 mg telotristat etiprate (LX1606) administered orally once daily (QD).
Arm/Group | Placebo | Low Dose LX1606 | High Dose Telotristat Etiprate
Number analyzed (Participants) | 10 | 24 | 24
participants | 3 | 9 | 10

2. Secondary Outcome: Number of Participants Achieving Clinical Response
Description: Clinical response is defined as a decrease in the total modified Mayo score from baseline of ≥3 or a ≥30% decrease in the total modified Mayo score from baseline, along with a decrease in the rectal bleeding score ≥1 or an absolute rectal bleeding score ≤1 at Week 8.
  A modified Mayo score was used to evaluate disease activity using 4 components, including stool frequency, rectal bleeding, endoscopy, and physician assessment. Components = Stool frequency score 0-3 (normal- >4 stools/day more than normal), rectal bleeding score 0-3 (none-passing blood alone), mucosal appearance at endoscopy 0-3 (normal-severe disease), physician rating of disease activity 0-3 (normal-severe). The total Modified Mayo score ranges from 0 to 12, with higher scores indicating greater disease severity.
Time Frame: Baseline to 8 weeks
Population: Intent-to-treat (ITT) Population included all randomly assigned participants.
Measure: Number; unit: participants
Arm/Group | Placebo | Low Dose Telotristat Etiprate | High Dose Telotristat Etiprate
Number analyzed (Participants) | 10 | 25 | 24
participants | 4 | 8 | 8

3. Secondary Outcome: Number of Participants Achieving Clinical Remission
Description: Clinical remission is defined as a total modified Mayo score ≤2 with no individual score >1 at Week 8.
  A modified Mayo score was used to evaluate disease activity using 4 components, including stool frequency, rectal bleeding, endoscopy, and physician assessment. Components = Stool frequency score 0-3 (normal- >4 stools/day more than normal), rectal bleeding score 0-3 (none-passing blood alone), mucosal appearance at endoscopy 0-3 (normal-severe disease), physician rating of disease activity 0-3 (normal-severe). The total Modified Mayo score ranges from 0 to 12, with higher scores indicating greater disease severity.
Time Frame: Baseline to 8 weeks
Population: ITT Population included all randomly assigned participants.
Measure: Number; unit: participants
Arm/Group | Placebo | Low Dose Telotristat Etiprate | High Dose Telotristat Etiprate
Number analyzed (Participants) | 10 | 25 | 24
participants | 2 | 2 | 3

4. Secondary Outcome: Change From Baseline in Total Modified Mayo Score
Description: A modified Mayo score was used to evaluate disease activity using 4 components, including stool frequency, rectal bleeding, endoscopy, and physician assessment. Components = Stool frequency score 0-3 (normal- >4 stools/day more than normal), rectal bleeding score 0-3 (none-passing blood alone), mucosal appearance at endoscopy 0-3 (normal-severe disease), physician rating of disease activity 0-3 (normal-severe). The total Modified Mayo score ranges from 0 to 12, with higher scores indicating greater disease severity.
Time Frame: Baseline to 8 weeks
Population: Participants from the ITT Population, all randomly assigned participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose Telotristat Etiprate | High Dose Telotristat Etiprate
Number analyzed (Participants) | 8 | 19 | 19
units on a scale | -2.38 (2.973) | -1.89 (2.865) | -2.53 (2.389)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo | Low Dose Telotristat Etiprate | High Dose Telotristat Etiprate
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/24 | 2/24
Other Adverse Events (participants affected / at risk) | 3/10 | 9/24 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Low Dose Telotristat Etiprate (N=24) | High Dose Telotristat Etiprate (N=24)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Low Dose Telotristat Etiprate (N=24) | High Dose Telotristat Etiprate (N=24)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least sixty (60) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any information to which Sponsor objects, any Confidential Information, proprietary information or patentable subject matter.